CLINICAL TRIAL: NCT00989859
Title: A Pilot Study Using Photo-plethysmographic (PPG) Camera to Monitor Heart Rate, Respiration Rate and Oxygen Saturation in Infants.
Brief Title: Photo-Plethysmographic Camera to Monitor Heart Rate, Respiration Rate and Oxygen Saturation in Infants
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Willem Verkruysse, Ph.D., Associate Specialist, University of California, Irvine
Other Study IDs: 20097046.
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Child Development
Keywords: monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Plethysmographic monitoring: Plethysmographic monitoring
  Interventions: Device: Plethysmographic monitoring

INTERVENTIONS:
Device: Plethysmographic monitoring — Plethysmographic monitoring

SUMMARY:
The researchers want to determine if ambient light, plethysmographic , can monitor reliably heart rate, respiration rate and oxygen saturation in infant patients in a hospital setting.

DETAILED DESCRIPTION:
The plethysmographic signal is typically strong on children. This provides a reliable heart rate monitor. However, to measure oxygen saturation, a quantitative value of the strength at two wavelength regions (green and red) is required. It is also not known if the normal ambient light is spectrally appropriate to analyze the video signals for oxygenation. With the current prototype of our system, we can monitor heart rate reliably and estimate oxygen saturation in adults, using normal artificial light or daylight, entering through a window. Heart rate and oxygen saturation will be extracted from the plethysmographic signal off the cheek, forehead or hand while the respiration rate may be retrieved from the plethysmographic signal off the chest area.

ELIGIBILITY:
Inclusion Criteria:

* infant in NICU at CHOC hospital

Exclusion Criteria:

* non-infant

Ages: 1 Minute to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infant
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
ambient light, PPG can monitor reliably heart rate, respiration rate and oxygen saturation (SpO2) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Nelson, MD, Study Director — Beckman Laser Institute University of California Irvine; William Verkruysse, PhD, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- CHOC, Orange, California, United States